MyMenoPlan: Online Resource for Improving Women's Menopause Knowledge and Informed Decision-making
NCT05299983
10 January 2022

## **Consent Form**

You are being invited to participate in a research study. The purpose of the study is to learn how well women's needs are met by websites about perimenopause and menopause. Your feedback will help us improve our site and learn how our website compares to other sites. This study is being done by Drs. Andrea Z. LaCroix (University of California San Diego), Leslie Snyder (University of Connecticut), and Katherine M. Newton (Kaiser Permanente Washington Health Research Institute).

If you agree to be in this study, we will ask you to explore a website for at least 20 minutes, and then complete a 15 minute questionnaire. The questionnaire will ask about your menopausal status, your menopause symptoms, and your reaction to the website, as well as your age, race/ethnicity, and education. You will receive a \$30 gift card 1-2 weeks after you complete the questionnaire as a token of appreciation for your participation.

You will be randomly assigned to one of two groups. One group will use a new website we developed. The other group will use another other website. If you are not assigned to see our website now, we can send you a link to the website after the study is over. The project team cannot change your group.

You are eligible to participate in the study if:

- 1. You are a woman 40 to 60 years old.
- 2. You have questions about perimenopause or menopause or you have at least one bothersome symptom.
- 3. You did not participate in the My Menoplan pilot study.

You may directly benefit from using these websites by learning more about perimenopause, menopause, symptoms, treatments, and coping strategies, and developing a personalized plan to manage your symptoms.

Your participation in this study is completely voluntary and you can withdraw at any time by simply exiting the survey. Choosing not to participate or withdrawing will result in no penalty or loss of benefits to which you are entitled. You are free to not answer any question that you choose.

To send you the gift card and verify your identity, we will collect some private information, including your name, email address, phone, and mailing address. Your computer's IP address will be used to match your website use to your questionnaire. (An IP address is a unique address that identifies your electronic device.)

## You will be disqualified from the study and not paid if you:

- do not meet the study eligibility criteria,
- do not review the assigned website for at least 20 minutes,
- do not complete the questionnaire,
- we cannot verify your identity.

These procedures help us prevent fraudulent study participation. Unfortunately, fraud is very common and can invalidate the study findings.

You may only participate once. Only one person per household may participate.

Research records will be kept confidential to the extent allowed by law and may be reviewed by the UCSD Institutional Review Board. There are minimal risks associated with this research study.

There is a small risk of breach of confidentiality of your private information. To minimize this risk, all private information will be kept in a password-protected file that is separate from your data. Private information will be destroyed when the study is complete. If you have any questions about the study or our website, you can call 860-341-2101. If you have questions about your rights as a research participant, you may contact the UC San Diego Human Research Protections Program Office at 858-246-4777. This program is a group of people who review research studies to protect the welfare of research participants.

By clicking "You agree" below you are indicating that you are at least 18 years old, have read this consent form, and agree to participate in this research study. (You may print a copy of this page for your records.)

| O You Agree (1) | |
|--------------------|-----|
| O You Do Not Agree | (2) |